CLINICAL TRIAL: NCT03386929
Title: A Proof of Concept Study to Explore Safety and Efficacy of Tri-therapy Approach in Advanced/Metastatic NSCLC and Retrospectively Assess the Ability of Integrated Genomics and Transcriptomics to Match Patients to the Combination
Brief Title: Survival Prolongation by Rationale Innovative Genomics
Acronym: SPRING
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The SPRING trial had to be early terminated at the end of the Phase 1 portion of the study due to the absence of funding necessary for the performance of the Phase 2.
Sponsor: Worldwide Innovative Network Association (Other)
Collaborators: ARC Foundation for Cancer Research (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIN001; 2017-001455-32 (EudraCT Number)
Record Dates: First submitted 2017-12-14; First posted 2017-12-29 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Non-small Cell Lung Cancer Stage IIIB
Keywords: NSCLC; tri-therapy; avelumab; axitinib; palbociclib; dual matched normal and tumor biopsies; SIMS algorithm; Sequencing; Gene expression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — avelumab; Axitinib; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab, Axitinib, Palbociclib (Experimental): For the Phase 1:
  Avelumab is administered intravenously (IV) on Day 1 and Day 15 of a 28 day cycle in combination with axitinib po bid (every day of a 28 day cycle) and palbociclib po (on days 8-28 of a 28 day cycle).
  For the Phase 2:
  Avelumab, axitinib and palbociclib are administered at the recommended phase 2 dose (RP2D) as determined during the phase 1 part of the study.
  Interventions: Drug: Avelumab; Drug: Axitinib; Drug: Palbociclib

INTERVENTIONS:
Drug: Avelumab — A human antibody of the immunoglobulin gamma-1 isotype that specifically targets and blocks the Programmed Death ligand (PD-L1) for PD-1.
Drug: Axitinib — A selective oral (tablet) inhibitor of tyrosine kinases Vascular Endothelial Growth Factor (VEGF) receptors 1, 2, and 3. These receptors are implicated in pathologic angiogenesis, tumor growth and cancer progression.
  Other Names: Inlyta
Drug: Palbociclib — A selective, reversible oral (capsule) inhibitor of cyclin-dependent kinases (CDK) 4 and 6. The inhibition of CDK 4/6 blocks DNA synthesis by prohibiting progression of the cell cycle from G1 to S phase.
  Other Names: Ibrance

SUMMARY:
Patients with advanced/metastatic non-small cell lung cancer (NSCLC) with no documented targetable alterations (Epidermal Growth Factor Receptor (EGFR) mutation, Anaplastic Lymphoma Kinase (ALK) translocation, ROS1 mutation if available or MET exon 14 skipping mutation if available) will receive a tri-therapy associating avelumab, axitinib and palbociclib.

DETAILED DESCRIPTION:
During the Phase 1 (approximately 30 patients), the tri-therapy will be tested at different doses following a specific dose-escalation scheme (3 + 3 model) in order to establish the safety and identify the Maximum Tolerated Dose (MTD) and recommended dose for the Phase 2 (RP2D). The phase 2 will confirm the safety and will assess the clinical utility of the tri-therapy approach in the treatment of advanced/metastatic NSCLC (100 patients). The study will also explore the clinical utility of the Simplified Interventional Mapping System (SIMS), a new tool/algorithm enabling matching of NSCLC patients with combination therapy. For this purpose tumor/metastasis and matched normal tissue biopsies will be requested in order to obtain sequencing and expression profiles.

ELIGIBILITY:
ELIGIBILITY CRITERIA

* Age: Men and women aged >18 years,
* Signed written informed consent,
* Any histologic type of locally advanced or metastatic NSCLC,
* Life expectancy of ≥ 12 weeks,
* Measurable or evaluable (cytologically or radiologically detectable disease such as ascites, peritoneal deposits, or lesions which do not fulfill RECIST 1.1 criteria for measurable disease) lesions according to RECIST 1.1 criteria for phase 1 portion. For phase 2, all patients must have RECIST 1.1 measurable disease,
* Physiologic function:

  * Hematologic: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused),
  * Hepatic: Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 × ULN,
  * Renal: Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).
* Pregnancy and contraception:

  * Pregnancy test: Negative serum or urine pregnancy test at screening for women of childbearing potential.
  * Contraception: Highly effective contraception for both male and female subjects throughout the study and for at least 90 days after last treatment administration if the risk of conception exists.
* Ability to comply with protocol requirements,
* Willingness to consent and ability to undergo a trucut biopsy to obtain a fresh metastasis or primary tumor biopsy, and to undergo bronchoscopy to obtain a biopsy from normal bronchial mucosa,
* No serious or medically uncontrolled concomitant conditions that are likely to make the patient unfit for SPRING combination therapy, as per investigator assessment,
* ECOG performance status of 0 to 1.

EXCLUSION CRITERIA

* Patients with documented oncogenic aberrations at enrollment: EGFR, ALK, ROS1 when available, MET exon 14 skipping when available. For squamous undifferentiated cell carcinoma, documentation of these aberrations is not mandatory. Note: For Phase 1 portion, all patients with adenocarcinoma histology must have documentation of results for druggable oncogenic aberrations (EGFR mutations, ALK rearrangements, and ROS1 when available) prior to enrollment on the study.
* For Phase 1 portion, >2 lines of prior therapy in the metastatic setting.
* For the dose escalation phase of the study or until the MTD for the combination regimen has been determined, patients with moderate hepatic impairment defined as AST, ALT, alkaline phosphatase (ALP) >5 times ULN, which would be grade 3 or higher. However, patients with liver metastases with AST/ALT ≤ 5 x ULN can be included in the study.
* For Phase 2 portion, any prior therapy in the metastatic setting.

Clinical criteria for phase 1 and phase 2 studies:

* Patients with treated brain metastases are eligible as are patients with new, active untreated brain metastasis.
* Participants with a history of myocardial infarction within the last 2 years or with significant cardiac arrhythmias uncontrolled by medication or pacemaker,
* Participants with any history of interstitial lung disease,
* Prior clinically significant toxicities from anticancer agents or radiotherapy which have not regressed to Grade ≤ 1 severity (NCI-CTCAE version 4.03) apart from peripheral neuropathy and alopecia,
* History of any second malignancy in the last two years; patients with prior history of in-situ cancer or basal or squamous cell skin cancer are eligible. Patients with a history of other malignancies are eligible if they have been continuously disease-free for at least two years,
* Autoimmune condition requiring medical intervention,
* Uncontrolled concomitant illness, active infection requiring i.v. antibiotics,
* Patients who have had a thromboembolic event within six months are excluded, as are patients on anticoagulants, except for low dose aspirin (<100 mg/day) and low doses of anticoagulants meant to keep line access open;
* Patients with Grade 3 or 4 (serious) gastrointestinal bleeding within the last six months are excluded.
* Prior > G3 hemoptysis, major blood vessel involvement (specifically including aorta, superior and inferior vena cave, main pulmonary arteries and veins, subclavian arteries and veins and other large blood vessels that in the investigator's opinion places the patients at high risk for major bleeding), and/or central cavitations,
* Known or suspected drug hypersensitivity to any drug used in the combination,
* Difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the oral drugs,
* Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location, etc.) that, in the judgment of the investigator may affect the patient's ability to sign the informed consent and undergo study procedures,
* Taking another experimental drug within 28 days prior to day 1 of the protocol medications in this study,
* Pregnant or breast-feeding women,
* Both male and female patients of reproductive potential must agree to use highly effective contraception, during the study and for 3 months following the last dose of study drug,
* Patients currently taking strong CYP3A4 inducers and inhibitors,
* Patients currently taking proton pump inhibitors due to their impact on the disposition of palbociclib during the phase 1.
* Patients taking other anticancer agents with the exception of denosumab or equivalent medication for bone metastases.
* A time period of at least three weeks (including radiotherapy) or five drug half-lives, whichever is shorter must have elapsed from last non-investigational therapy before first day of treatment on this study,
* A time period of at least 10 days must have elapsed from last palliative radiotherapy before the first day of treatment on this study,
* Specific exclusion criteria for administration of avelumab, in combination:

  * IMMUNOSUPRESSANTS: Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
  * AUTOIMMUNE DISEASE: Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
  * ORGAN TRANSPLANTATION: Prior organ transplantation including allogenic stem-cell transplantation.
  * INFECTIONS: Active infection requiring IV (Intra venous) therapy.
  * HIV/AIDS: Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
  * HEPATITIS: Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
  * VACCINATION: Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
  * HYPERSENSITIVITY TO STUDY DRUG: Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
  * CARDIOVASCULAR DISEASE: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia inadequately controlled by medication.
  * OTHER PERSISTING TOXICITIES: Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
  * Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: RAZELLE KURZROCK, MD, Principal Investigator — Medical College of Wisconsin, Milwaukee, WI, USA
Locations (5):
- United States (2):
  - UCSD Moores Cancer Center, La Jolla, California
  - Avera Cancer Center, Sioux Falls, South Dakota
- Chaim Sheba Medical Center, Ramat Gan, Israel
- Centre Hospitalier Luxembourg, Luxembourg, Luxembourg
- Vall Hebron Institute of Oncology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solomon B, Callejo A, Bar J, Berchem G, Bazhenova L, Saintigny P, Wunder F, Raynaud J, Girard N, Lee JJ, Sulaiman R, Prouse B, Bresson C, Ventura H, Magidi S, Rubin E, Young B, Onn A, Leyland-Jones B, Schilsky RL, Lazar V, Felip E, Kurzrock R. A WIN Consortium phase I study exploring avelumab, palbociclib, and axitinib in advanced non-small cell lung cancer. Cancer Med. 2022 Jul;11(14):2790-2800. doi: 10.1002/cam4.4635. Epub 2022 Mar 20. PMID 35307972
- See also: sponsor website — https://www.winconsortium.org/
- See also: SIMS article link: A simplified interventional mapping system (SIMS) for the selection of combinations of targeted treatments in non-small cell lung cancer. — http://www.oncotarget.com/index.php?journal=oncotarget&page=article&op=view&path[]=3741&pubmed-linkout=1
- See also: Link to the publication of the results of the Phase 1 part of the study — https://pubmed.ncbi.nlm.nih.gov/35307972/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 patients were recruited in the Phase 1 part of the study in 5 centers across 4 countries (Luxembourg, Israel, Spain and USA). The study was early terminated prior starting the Phase 2 due to lack of fundings.
  The following number of treated patients were initially planned to be recruited:
  up to 30 in the Phase 1 and 100 in the Phase 2.
Pre-assignment Details: Patients with advanced/metastatic advanced/metastatic non-small cell lung cancer (NSCLC) with no documented targetable alterations (EGFR mutation, ALK translocation, ROS1 mutation if available or MET exon 14 skipping mutation if available) were recruited in the study.
Groups:
- Dose Level 1: Non-small cell lung cancer (NSCLC) patients treated with avelumab (10 mg/kg IV every two weeks -1/+3 days, on day 1 and day 15 of a 28 day cycle), axitinib (3 mg taken orally twice a day, every day of a 28 day cycle) and palbociclib (75 mg taken orally, daily on days 8-28 of a 28 day cycle).
- Dose Level 2: Non-small cell lung cancer (NSCLC) patients treated with avelumab (10 mg/kg IV every two weeks -1/+3 days, on day 1 and day 15 of a 28 day cycle), axitinib (5 mg taken orally twice a day, every day of a 28 day cycle) and palbociclib (75 mg taken orally, daily on days 8-28 of a 28 day cycle).
- Dose Level 3: Non-small cell lung cancer (NSCLC) patients treated with avelumab (10 mg/kg IV every two weeks -1/+3 days, on day 1 and day 15 of a 28 day cycle), axitinib (5 mg taken orally twice a day, every day of a 28 day cycle) and palbociclib (100 mg taken orally, daily on days 8-28 of a 28 day cycle).
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 6 | 6 | 3
Completed | 0 | 0 | 0
Not Completed | 6 | 6 | 3
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Progression | 4 | 4 | 0
Not completed — Clinical Monitoring Committee and physician choice | 1 | 1 | 1
Not completed — Transfer to SPRING Rollover protocol (EU CT # 2022-500041-24-00) after closing SPRING | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 6 | 6 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 2 | 7
  >=65 years | 3 | 4 | 1 | 8
Age, Continuous [Median (Full Range); unit: years] | 68 [52 to 80] | 67 [51 to 72] | 54 [51 to 76] | 67 [51 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 5
  Male | 3 | 5 | 2 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 6 | 2 | 14
  Mexican | 0 | 0 | 1 | 1
  Black | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 0 | 2 | 7
  Luxembourg | 0 | 2 | 0 | 2
  Israel | 0 | 2 | 1 | 3
  Spain | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of the Tested 3-Drug Combination Therapy-Emergent Adverse Events and Serious Adverse Events
Description: The occurrence of adverse events and serious adverse events reported from the signing of an informed consent through 90 days after the last administration of the treatment will be summarized for all subjects who received at least one dose of the study treatment (safety population) and will be evaluated based on NCI CTCAE v4.03: June 14, 2010.
Time Frame: From informed consent signature through 90 days after administration of the treatment (last dose)
Population: This outcome could not be measured because the data were not collected. Indeed, the trial was early terminated after the end of the phase 1. The phase 2 was not started, no data can be reported.
Groups:
- Planned Population for Analysis: 100 treated patients in the Phase 2 including patients enrolled in the Phase 1 at the recommended Phase 2 dose. The planned population for analysis of response (evaluable patients) was those that received at least one cycle of treatment.
Arm/Group | Planned Population for Analysis
Number analyzed (Participants) | 0

2. Primary Outcome: Response Rate (RR)
Description: Response rate is defined as the proportion of participants with reduction in tumor burden of a predefined amount based on RECIST 1.1 evaluation
Time Frame: Baseline up to approximately 24 months
Population: as for outcome 1
Arm/Group | Planned Population for Analysis
Number analyzed (Participants) | 0

3. Primary Outcome: Duration of the Response
Description: Duration of Response (DR) is defined for patients with confirmed objective response (Complete Response [CR] or Partial Response [PR]) as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Time Frame: Baseline up to approximately 24 months
Population: as for outcome 1
Arm/Group | Planned Population for Analysis
Number analyzed (Participants) | 0

4. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression Free Survival (PFS) is defined as the time from the first dose of study treatment to the date of disease progression by RECIST 1.1 or death due to any cause, whichever occurs first.
Time Frame: Baseline up to approximately 24 months
Population: as for outcome 1
Arm/Group | Planned Population for Analysis
Number analyzed (Participants) | 0

5. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first dose of study treatment to the date of death due to any cause.
Time Frame: Baseline up to approximately 24 months
Population: as for outcome 1
Arm/Group | Planned Population for Analysis
Number analyzed (Participants) | 0

6. Primary Outcome: SIMS Algorithm to Predict Clinical Outcome
Description: The proportion of participants whose SIMS analysis matches the treatment combination, will be correlated retrospectively to clinical outcome.
Time Frame: 4 years
Population: as for outcome 1
Arm/Group | Planned Population for Analysis
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of Treatment-related and or Biopsy-related Serious Adverse Events
Description: The occurrence of treatment-related and or biopsy-related serious adverse events as assessed by NCI CTCAE v4.03 will be summarized for all study subjects.
Time Frame: 4 years
Population: as for outcome 1
Arm/Group | Planned Population for Analysis
Number analyzed (Participants) | 0

8. Secondary Outcome: Genomic and Transcriptomic Profile
Description: Genomic (DNA) and transcriptomic (RNA) aberrations (mutations, translocations, rearrangements and changes in expression level) identified in the study population (Non-Small Cell Lung) will be described.
Time Frame: 4 years
Population: as for outcome 1
Arm/Group | Planned Population for Analysis
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the time of Informed Consent through the follow-up period of 90 days after discontinuation of the study treatment, up to 4,5 years.
Description: AEs were graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
  Causal relationship between study treatment and AEs was determined by the investigators and the clinical monitoring committee, and events were considered drug-related if classified by the investigator as at least possibly related to study treatment.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/6 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/6 | 2/3
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=6) | Dose Level 3 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=6) | Dose Level 3 (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (9) | 3 (5) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (3) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (4) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (11) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Temperature regulation disorder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Urinary Tract infection (Infections and infestations) | 1 (2) | 1 (6) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 5 (13) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 2 (4) | 2 (3) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase increased (Investigations) | 0 (0) | 2 (4) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (4) | 3 (10) | 1 (2)
Neutrophil count decreased (Investigations) | 4 (28) | 3 (8) | 0 (0)
Platelet count decreased (Investigations) | 3 (7) | 4 (14) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 2 (4) | 1 (1)
White blood cell count decreased (Investigations) | 4 (13) | 3 (7) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (9) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (12) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (6) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (6) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (5) | 1 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (12) | 2 (5) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail Ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (6) | 4 (11) | 3 (3)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was early terminated after the end of its Phase 1 due to lack of funding. As a result it was not possible to analyse the objectives of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03386929/Prot_SAP_000.pdf